CLINICAL TRIAL: NCT04929847
Title: Evaluation of a Novel Skin Care Product for the Management of Chemotherapy- Related Dermatologic Toxicities
Brief Title: Novel Skin Care for Chemotherapy- Related Dermatologic Toxicities
Acronym: ChemoSkin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jessa Hospital (Other)
Collaborators: Hasselt University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021/060
Record Dates: First submitted 2021-06-11; First posted 2021-06-18 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Skin Toxicity
Keywords: chemotherapy; skin; emollient; oncology
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group 1 (Experimental): All patients will receive the experimental emollient during 3 weeks.
  Interventions: Other: Self-prepared emollient

INTERVENTIONS:
Other: Self-prepared emollient — The emollient is hypo-allergenic, free of perfume and has very high hydrating capacities together with antioxidants.

SUMMARY:
Notwithstanding the continuous progress in cancer treatment, patients with cancer still have to cope with quality of life (QoL) - impairing complications. Especially an extensive spectrum of dermatologic toxicities has been associated with cancer treatments. The number and type of cutaneous toxicities have evolved over the past 50 years, paralleling the development of new chemotherapeutic agents. The chemotherapy-related skin toxicities can significantly impede the patient's emotional, physical, social, and financial well-being resulting in a poor QoL. In rare cases of severe cutaneous reactions, treatment modifications are needed, resulting in a diminished overall survival.

Important organizations in the field of oncology and supportive care, such as the MASCC, the ASCO, and the ESMO, have developed guidelines for the management of cancer therapy- related cutaneous toxicities based on available scientific evidence. Still, for some interventions, the evidence of recommendation is moderate to insufficient. Therefore, it is essential to elucidate other new potential management strategies for dermatological complications of cancer treatment. Based on the previously mentioned supportive care guidelines for the ChemoSkin project, a novel emollient to tackle the cutaneous adverse events of chemotherapy has been developed.

The ChemoSkin project general aim is to evaluate the efficacy of a novel skincare product to manage chemotherapy-related cutaneous toxicities.

DETAILED DESCRIPTION:
Primary objective Evaluate the efficacy of a novel emollient for the management of chemotherapy-related cutaneous adverse events

Secondary objective 1 Evaluate patient-relevant treatment benefit of the novel emollient for chemotherapy-associated cutaneous toxicities

Secondary objective 2 Evaluate the influence of the novel emollient for chemotherapy- associated cutaneous toxicities on the patient's quality of life

Secondary objective 3 Evaluate the safety of the novel emollient for chemotherapy- associated cutaneous toxicities

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with cancer of any type
* Undergoing chemotherapy at the Jessa Hospital (Hasselt, BE)
* Age ≥ 18 years
* Able to comply to the study protocol
* Able to sign written informed consent

Exclusion Criteria:

* Pre-existing skin rash, ulceration, skin infections or open wounds
* Severe psychological disorder or dementia
* Any condition that is unstable or could affect the safety of the patient and their compliance in the study as judged by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-10-20 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Skin reaction evaluation | Baseline
  The severity of the skin reactions will be evaluated by the National Cancer Institute-Common Terminology Criteria for Adverse Events version 5 (NCI-CTCAE v5.
Skin reaction evaluation | Week 3 of chemotherapy (End of study)
  The severity of the skin reactions will be evaluated by the National Cancer Institute-Common Terminology Criteria for Adverse Events version 5 (NCI-CTCAE v5.
Patient benefit composite | Baseline
  The Patient Benefit Index is a standardized questionnaire measuring patients' treatment needs and treatment benefits for skin diseases. The PBI comprises two components:
  1. Patient Needs Questionnaire measuring the importance of different treatment goals from the patient perspective.
  2. Patient Benefit Questionnaire measuring the achievement of the treatment goals from the patient perspective.
Patient benefit composite | Week 3 of chemotherapy (end of study)
  The Patient Benefit Index is a standardized questionnaire measuring patients' treatment needs and treatment benefits for skin diseases. The PBI comprises two components:
  1. Patient Needs Questionnaire measuring the importance of different treatment goals from the patient perspective.
  2. Patient Benefit Questionnaire measuring the achievement of the treatment goals from the patient perspective.

SECONDARY OUTCOMES:
Patient subjective evaluation of skin reactions | Baseline
  The patients will be asked to complete a questionnaire to evaluate the intensity of five common symptoms of skin reactions: pruritus, dryness, erythema, burning sensation, and pain on an 11-point Numerical Rating Scale
Patient subjective evaluation of skin reactions | Week 1 of chemotherapy
  The patients will be asked to complete a questionnaire to evaluate the intensity of five common symptoms of skin reactions: pruritus, dryness, erythema, burning sensation, and pain on an 11-point Numerical Rating Scale
Patient subjective evaluation of skin reactions | Week 2 of chemotherapy
  The patients will be asked to complete a questionnaire to evaluate the intensity of five common symptoms of skin reactions: pruritus, dryness, erythema, burning sensation, and pain on an 11-point Numerical Rating Scale
Patient subjective evaluation of skin reactions | Week 3 of chemotherapy (end of study)
  The patients will be asked to complete a questionnaire to evaluate the intensity of five common symptoms of skin reactions: pruritus, dryness, erythema, burning sensation, and pain on an 11-point Numerical Rating Scale
Quality of life - DLQI | Baseline
  Dermatology Life Quality Index (DLQI) is a questionnaire with 10 items and is used to measure QoL of dermatological patients.
Quality of life - DLQI | Week 3 of chemotherapy (end of study)
  Dermatology Life Quality Index (DLQI) is a questionnaire with 10 items and is used to measure QoL of dermatological patients.
Quality of life - Skindex-29 | baseline
  The skindex-29 is a validated instrument to measures patients' QoL specifically correlated with skin conditions. It has 3 scales addressing emotions (10 items), symptoms (7 items) and functioning (12 items).
Quality of life - Skindex-29 | Week 3 of chemotherapy (end of study)
  The skindex-29 is a validated instrument to measures patients' QoL specifically correlated with skin conditions. It has 3 scales addressing emotions (10 items), symptoms (7 items) and functioning (12 items).
Patients' satisfaction with the therapeutic intervention | Week 3 of chemotherapy (end of study)
  The patients will be asked to evaluate the general pleasantness and soothing effect of the skin care products by using a numerical rating scale.

OTHER OUTCOMES:
General patient-, disease-, and treatment-related information | Baseline
  General and medical information will be collected through a short patient questionnaire in order to assess intrinsic risk factors (i.e., gender, age, smoking history, work habits, physical activity, skin condition, alcohol use, and medication use). Furthermore, information about disease- and treatment-related risk factors will be collected through medical records (e.g., tumor type and stage, tumor site, treatment type, radiotherapy regimen).

CONTACTS AND LOCATIONS:
Overall Officials: Jeroen Mebis, MD, PhD, Principal Investigator — Jessa Ziekenhuis VZW
Locations (1):
- Jessa Ziekenhuis VZW, Hasselt, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Manuscript: "Evaluation of a novel skin care product for the management of chemotherapy- related dermatologic toxicities: A quasi-experimental study" — https://doi.org/10.1016/j.ejon.2023.102278